CLINICAL TRIAL: NCT04687852
Title: Comparison of the Efficacy of Pharmacology and Non-pharmacological Treatment in Women With Primary Dysmenorrhea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.66761
Record Dates: First submitted 2020-12-10; First posted 2020-12-29 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-06

CONDITIONS: Pelvic Floor; Exercise; Telerehabilitation; Acupressure; Dysmenorrhea Primary; Drug Effect
Keywords: Pelvic Floor; Dysmenorrhea Primary; Drug therapy; Telerehabilitation; Acupressure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Focused Pelvic Floor Exercise with Motor ImageryTechnique Group (Experimental): 5 minute-Meditation Therapy 10 minute-Progressive Relaxation training ( Bernstein-Borkovec Method) 5 min - Breathing Exercises (Diaphragmatic Breathing Exercise, Pursed lip breathing Exercise) 35 min -Motor Imagery Technique Focused Pelvic Floor Exercises-MOPEXE 5 min - Meditation Therapy Twice a week for 60 minutes 12 weeks Participants will be evaluated online at the beginning of the research and at the end of the 12-week program.
  Interventions: Other: Conservative and Non-conservative treatments
- Nonsteroidal Anti-Inflammatory Drug(NSAID) Group (Active Comparator): Naproxen Sodium 550 mg film-coated tablet prescribed by the physician will be given to patients. During the menstrual period, 1 or 2 times a day will be used depending on the pain of the patient. Treatment time; 12 weeks.
  Interventions: Other: Conservative and Non-conservative treatments
- Diosmin Group (Other): Diosmin (90%) 500 mg film-coated tablets prescribed by the physician will be given to patients. During the menstrual period, 1 or 2 times a day will be used depending on the patient's pain. Treatment time; 12 weeks.
  Interventions: Other: Conservative and Non-conservative treatments
- Acupressure Group (Experimental): 4 acupuncture points will be applied twice a day for 12 weeks. These points are; LI4, CV4, CV6, SP6
  .
  Interventions: Other: Conservative and Non-conservative treatments
- Control Group (No Intervention): Participants will not be treated.

INTERVENTIONS:
Other: Conservative and Non-conservative treatments — This program includes Focused Pelvic Floor with Motor Imagery Technique Group ,Nonsteroidal Anti-Inflammatory Drug Group, Diosmin Group, Acupressure Group (LI-4 (Bilateral), CV-6, CV-4, SP-6 (Bilateral). It is aimed to determine the most effective treatment among these groups.
  Arms: Acupressure Group; Diosmin Group; Focused Pelvic Floor Exercise with Motor ImageryTechnique Group; Nonsteroidal Anti-Inflammatory Drug(NSAID) Group

SUMMARY:
Primary dysmenorrhea is a common problem in women. Women use many treatment methods to deal with primary dysmenorrhea. Therefore, this study aims to find the most effective treatment by determining the effectiveness of conservative and non-conservative treatment in women with primary dysmenorrhea. Another aim of the study is to generalize the use of conservative treatment methods in the treatment of primary dysmenorrhea.On the other hand, it aims to spread the telerehabilitation method, which allows the global Covid 19 outbreak to be maintained remotely online, in the world and in our country.

DETAILED DESCRIPTION:
This study aims to determine the effects of different treatment approaches in women diagnosed with primary dysmenorrhea. Patients who are examined by a physician and diagnosed with primary dysmenorrhea using ultrasonography will be included in the study. The cases will be divided into 5 groups by randomization. In the first group, patients who are prescribed diosmin by the attending physician will be taken. The second group; Patients who are prescribed naproxen sodium by the attending physician will be taken. The third group; Pelvic floor exercises will be performed 2 days a week and 12 weeks a week using the motor imagination technique created by the women health physiotherapist. In the fourth group, acupressure technique applied by applying pressure to non-invasive acupuncture points will be applied daily for 12 weeks. The fifth group will be the control group. Online access will be synchronized with the phone or computer, and training sessions will not be recorded to protect the patient's personal information. Cases will be evaluated online at the beginning of the study and at the end of the 12-week program.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 whose menstrual cycle continues,
* Primary dysmenorrhea was diagnosed by the obstetrician by ultrasonographic evaluation.
* Participants who agree to participate in the study will be included.
* Participants in the diosmin group who were prescribed diosmin by the physician
* Participants in the NSAI group who were prescribed an NSAI by the physician

Exclusion Criteria:

* Receiving hormone therapy
* Those receiving psychiatric treatment for stress disorder or anxiety
* Intrauterine contraceptive device
* Using birth control pills
* Women diagnosed with secondary dysmenorrhea
* With neurological deficits
* Patients who were not suitable for NSAI and Diosmin treatment by the physician were excluded by the physician and were not included in our study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | 5 minutes
  Participants age, height, weight, educational status, marital status, exercise habits will be recorded. In addition, sociodemographic information, clinical features such as background and family history; Information on menarche age, average cycle duration and menstruation duration, and methods of coping with dysmenorrhea were recorded.
Visual Analogue Scale (VAS) | 2 minutes
  The Visual Analogue Scale (VAS) is used to convert non-numerical values to digital. The value 0 means I have no pain, 10 means I have unbearable pain. The person marks his pain on this ruler. It measures the intensity of the pain.
McGill Pain Questionnaire | 5 minutes
  The characteristic of pain felt by the patients during menstruation was evaluated using the McGill Pain Questionnaire-Short Form,With the McGill Melzack Pain Questionnaire, the location of the pain, the feeling it creates in the individual, its relationship with time, its severity and the level of viable pain for the individual are determined. High score indicates high level of pain
Ultrasonography (US) | 5 minutes
  Ultrasonography is a soft tissue examination method.Its biggest advantages are that it is an easily accessible method and does not contain ionizing radiation.
  In the evaluation by ultrasonography, dysmenorrhea due to organic problems will be evaluated and excluded by the obstetrician.

SECONDARY OUTCOMES:
Menstrual Attitude Questionnaire | 5 minutes
  The Turkish version of the Menstrual Attitude Scale (MBI) will be applied to determine the attitudes and behaviors of the participants during the menstrual period. Menstruation attitude scale includes 5 subtitles. These subheadings are;
  1. Menstruation as a debilitating event
  2. Menstruation as a bothersome event
  3. Menstruation as a natural event
  4. Ancipitation and prediction of the onset of menstruation
  5. Denial of any effect of menstruation

CONTACTS AND LOCATIONS:
Overall Officials: Gizem BOZTAŞ ELVERİŞLİ, Phd, Study Director — Istanbul Medipol Üniversitesi
Locations (1):
- Gizem BOZTAŞ, Istanbul, Kavacık, Turkey (Türkiye)